CLINICAL TRIAL: NCT02294890
Title: Does Fibrosis Diathesis Influence the Recovery of Knee Mobility After Total Knee Replacement?
Brief Title: Knee Stiffness in Fibrosis Diathesis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital Pellenberg (Other)
Responsible Party: Principal Investigator, Maarten Van Nuffel, Fellow, University Hospital Pellenberg
Other Study IDs: UHPellenberg
Record Dates: First submitted 2014-11-05; First posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Knee Replacement Arthroplasty; Fibrosis; Dupuytren's Disease
MeSH Terms: conditions — Fibrosis; Dupuytren Contracture | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Fibrosis diathesis: all patients will be checked for signs of fibrosis diathesis. This will be done by examining their hands for Dupuytren's nodules and contractures and recording risk factors associated with increased severity and risk of recurrence of Dupuytren's contracture. These include family history, bilateral DD, and ectopic lesions, age of onset less than 50 years, male gender, Ledderhose disease, first ray involvement, multiple ray involvement and ectopic fibromatosis.
  This way, two groups of patients will be identified: those with and those without signs of fibrosis diathesis.
  Interventions: Procedure: Total knee arthroplasty
- No fibrosis diathesis: all patients will be checked for signs of fibrosis diathesis. This will be done by examining their hands for Dupuytren's nodules and contractures and recording risk factors associated with increased severity and risk of recurrence of Dupuytren's contracture. These include family history, bilateral DD, and ectopic lesions, age of onset less than 50 years, male gender, Ledderhose disease, first ray involvement, multiple ray involvement and ectopic fibromatosis.
  This way, two groups of patients will be identified: those with and those without signs of fibrosis diathesis.
  Interventions: Procedure: Total knee arthroplasty

INTERVENTIONS:
Procedure: Total knee arthroplasty

SUMMARY:
At the standard follow-up moment one year after primary TKA for gonarthrosis, all patients will be checked for signs of fibrosis diathesis. This will be done by examining their hands for Dupuytren's nodules and contractures and recording risk factors associated with increased severity and risk of recurrence of Dupuytren's contracture. These include family history, bilateral DD, and ectopic lesions, age of onset less than 50 years, male gender, Ledderhose disease, first ray involvement, multiple ray involvement and ectopic fibromatosis.

This way, two groups of patients will be identified: those with and those without signs of fibrosis diathesis. For both groups, the range of motion (ROM) of the operated knee at 3 and 6 months will be retrieved in the charts, the ROM at 12 months will be measured at that time. Also, additional procedures performed to increase ROM postoperatively will be retrieved from the charts (e.g. continuous passive motion, mobilization under anesthesia). Other causes for knee stiffness will have to be recorded, since these will be the most important exclusion criteria.

In the patients with clear signs of finger contractures, any impression of increase of contracture over the past 12 months will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a total knee replacement for primary gonarthrosis with a minimum follow-up of 1 year

Exclusion Criteria:

* Patients undergoing a TKA for other reasons than primary gonarthrosis, e.g. after infection, posttraumatic arthritis,hemophilia,…
* Patients who had other problems after their TKA resulting in knee stiffness, e.g. infection, bleeding,…

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who undergo a total knee arthroplasty for primary gonarthrosis at a minimal age of 50 years showing signs of fibrosis diathesis at presentation can be included. Patients who do not show signs of fibrosis diathesis will serve as a control group.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Range of movement of the operated knee at 12 months postoperatively | 12 months
Additional procedures/interventions to gain motion | 12 months

SECONDARY OUTCOMES:
- Increase of contracture or appearance of the nodules and contractures in the hand after the knee surgery. | 12 months
KSS score for knee function | 12 months

REFERENCES:
- [Background] Abe Y, Rokkaku T, Ofuchi S, Tokunaga S, Takahashi K, Moriya H. An objective method to evaluate the risk of recurrence and extension of Dupuytren's disease. J Hand Surg Br. 2004 Oct;29(5):427-30. doi: 10.1016/j.jhsb.2004.06.004. PMID 15336743
- [Background] Hindocha S, Stanley JK, Watson S, Bayat A. Dupuytren's diathesis revisited: Evaluation of prognostic indicators for risk of disease recurrence. J Hand Surg Am. 2006 Dec;31(10):1626-34. doi: 10.1016/j.jhsa.2006.09.006. PMID 17145383
- [Background] Issa K, Rifai A, Boylan MR, Pourtaheri S, McInerney VK, Mont MA. Do various factors affect the frequency of manipulation under anesthesia after primary total knee arthroplasty? Clin Orthop Relat Res. 2015 Jan;473(1):143-7. doi: 10.1007/s11999-014-3772-x. PMID 25002219
- [Background] Lungu E, Desmeules F, Dionne CE, Belzile EL, Vendittoli PA. Prediction of poor outcomes six months following total knee arthroplasty in patients awaiting surgery. BMC Musculoskelet Disord. 2014 Sep 8;15:299. doi: 10.1186/1471-2474-15-299. PMID 25201448
- [Background] Smith SP, Devaraj VS, Bunker TD. The association between frozen shoulder and Dupuytren's disease. J Shoulder Elbow Surg. 2001 Mar-Apr;10(2):149-51. doi: 10.1067/mse.2001.112883. PMID 11307078